CLINICAL TRIAL: NCT07072507
Title: The Effect of Childbirth Preparation Classes on Spousal Support, Birth Preference, Birth Memory, and Birth Satisfaction
Brief Title: Childbirth Education Classes, Spousal Support, Birth Memory, Choice of the Birth Method, and Birth Satisfaction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Gonca Buran, Asosc. Prof., Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 10/29
Record Dates: First submitted 2025-06-27; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Birth; Education; Pregnancy; Birth Memory; Birth Satisfaction
Keywords: Childbirth Education Classes; Partner Support; Birth Memory; Birth Satisfaction; choice of the birth method

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to the non-spouse education group, the together spouse education group, and the clinic's usual care control group by simple randomization.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kontrol (No Intervention): Participants in the control group will not receive any intervention. They will be left to the clinic's usual care.
- Education Group (Experimental): The training group will be divided into two categories: a partnerless education group and a partnered education group. Participants will receive 2 hours of weekly childbirth preparation training over the course of five weeks.
  Interventions: Behavioral: Chilbirth Education

INTERVENTIONS:
Behavioral: Chilbirth Education — Participants divided into training groups will receive training on pregnancy, birth, breastfeeding, preparation for parenthood, and baby care in groups of 6-8 people, 2 hours a week for five weeks.
  Arms: Education Group

SUMMARY:
The research questions of this study are listed below.

1. Is the mean spouse support score of pregnant women who attend childbirth preparation education with their spouses higher than that of women in the group with unique participation in childbirth preparation education and the control group who were left to usual care?
2. Is the mean birth satisfaction scale score of pregnant women who attend childbirth preparation education with their spouses higher than that of women in the group with unique participation in childbirth preparation education and the control group who were left to usual care?
3. Is the mean birth memory and recall scale score of pregnant women who attend childbirth preparation education with their spouses higher than that of women in the group with unique participation in childbirth preparation education and the control group who were left to usual care?
4. Are the birth preferences of pregnant women who attend childbirth preparation education with their spouses significantly different from those of women in the group with unique participation in childbirth prep

DETAILED DESCRIPTION:
Pregnancy is a physiological process that can create significant physical, psychological, and emotional stress for women. During this time, they may experience various symptoms and complaints. The outcomes of pregnancy can be unpredictable, which is why it's crucial for pregnant women to receive ample support from those around them, particularly their spouses. As a result, many women may choose to attend prenatal preparation courses. Ultimately, every woman desires a safe and uncomplicated birth, tailored to her preferences, and with a high level of satisfaction.

The purpose of this randomized controlled experimental study is to determine the effect of childbirth preparation classes on perception of spouse support and birth satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Being able to speak and write Turkish
* Nulliparous
* Being in 30-32 weeks of pregnancy
* Having a singleton pregnancy

Exclusion Criteria:

* Having communication and psychological problems
* Having multiple pregnancies
* Being overweight and obese
* Being divorced or having lost a spouse
* Not attending more than one session of childbirth preparation classes with/without a spouse
* Filling out incomplete forms

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Physiologically, pregnancy occurs with the female gender.
Enrollment: 93 (Estimated)
Dates: Start 2025-06-28 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Introduction form | During registration (first day)
  Participants will complete a five-question introduction form, including four sociodemographic questions and a question about birth preferences.
Pre Education-Spousal Support During Pregnancy | During registration (first day)
  The Perception of Spousal Support in Pregnancy Scale (PSSPS) (22 questions) will be administered during registration. The lowest possible score from the total scale is 16, and the highest score is 80. High scores from the scale indicate that perceived spousal support during pregnancy is high, while low scores indicate that perceived spousal support is low.
After Education - Spousal Support During Pregnancy | After education (When Childbirth Education is Finish)
  The Perception of Spousal Support During Pregnancy Scale (PSSPS) (22 questions) will be administered after childbirth education . The lowest possible score from the total scale is 16, and the highest score is 80. High scores from the scale indicate high perceived spousal support during pregnancy, while low scores indicate low perceived spousal support.
Postpartum- Memories and Recall | First week postpartum (during first clinical check-up)
  Birth memories and how he remembered his birth will be assessed with the "Birth Memories and Recall Questionnaire (BirthMARQ)" The scale has six sub-dimensions, and each sub-dimension is scored on its own. It is a 7-point Likert scale.
  Emotional memory sub-dimension: High scores in this dimension indicate having negative feelings about the birth experience.
  Ambiguous Emotional Memory Sub-dimension: High scores in this dimension indicate having more ambiguous feelings about the birth experience.
  Centrality of memory sub-dimension: High scores indicate that the birth memory is more centralized in the mother.
  Consistency and reliving sub-dimension: High scores in this dimension indicate a more consistent birth memory and more reliving.
  Sensory memory sub-scale: Higher scores indicate increased sensory memory of the birth experience.
  Involuntary recall sub-scale: Higher scores indicate more frequent involuntary recall.
Postpartum-Birth Satisfaction Scale Short Form (BSE-S) | First week postpartum (during first clinical check-up)
  The Birth Satisfaction Scale Short Form (BSE-S), which uses a 5-point Likert scale, will be utilized to measure birth satisfaction. The scale ranges from a lowest score of 0 to a highest score of 40 points. As the score increases, so does the level of satisfaction. For this study, the cut-off scores have been divided into three equal parts as follows:
  * Low satisfaction level: less than 13 points
  * Medium satisfaction level: 14 to 27 points
  * High satisfaction level: 28 points or more

SECONDARY OUTCOMES:
Birth method preference | During registration (first day)
  A question will be used to measure birth method preference. Options;
  * Vaginal birth
  * Vaginal birth with epidural anesthesia
  * Cesarean birth with spinal anesthesia
  * Cesarean birth with general anesthesia
Childbirth method | First week postpartum (during first clinical check-up)
  The participant will be asked to report the childbirth method that took place.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludag University, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Personal data can be shared only with the consent of the individuals involved. It can be shared if the participants have sharing approval.

REFERENCES:
- [Background] Zamani P, Ziaie T, Lakeh NM, Leili EK. The correlation between perceived social support and childbirth experience in pregnant women. Midwifery. 2019 Aug;75:146-151. doi: 10.1016/j.midw.2019.05.002. Epub 2019 May 6. PMID 31125906
- [Background] Arisukwu O, Igbolekwu CO, Oyekola IA, Oyeyipo EJ, Asamu FF, Osueke ON. Spousal support during pregnancy in the Nigerian rural context: a mixed methods study. BMC Pregnancy Childbirth. 2021 Nov 15;21(1):772. doi: 10.1186/s12884-021-04135-3. PMID 34781883